CLINICAL TRIAL: NCT01051960
Title: Exercise Induced Pulmonary Hypertension in Systemic Sclerosis and Treatment With Ambrisentan: A Prospective Single Center, Open Label, Pilot Study
Brief Title: Exercise Induced Pulmonary Hypertension in Systemic Sclerosis and Treatment With Ambrisentan
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-000567
Record Dates: First submitted 2010-01-19; First posted 2010-01-20 (Estimated); Results first posted 2020-11-02 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Systemic Sclerosis; Shortness of Breath; Pulmonary Hypertension
Keywords: Systemic Sclerosis; connective tissue disease; Shortness of breath; Pulmonary Hypertension
MeSH Terms: conditions — Scleroderma, Systemic; Dyspnea; Hypertension, Pulmonary; Connective Tissue Diseases | interventions — ambrisentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ambrisentan (Experimental): ambrisentan dosed at either 5mg or 10mg orally once per day
  Interventions: Drug: Ambrisentan

INTERVENTIONS:
Drug: Ambrisentan — Ambrisentan 5mg or 10mg once daily
  Other Names: Letairis

SUMMARY:
The purpose of this study is to determine the clinical characteristics and hemodynamic profiles that predict exercise induced pulmonary hypertension in 15 patients with systemic sclerosis. The study also aims to determine the effectiveness of Ambrisentan for subjects with exercise induced Pulmonary Arterial Hypertension (PAH) with scleroderma

DETAILED DESCRIPTION:
The current literature addresses therapies for patients with resting PAH only, diagnosed by right heart catheterization. However, the World Health Organization (WHO) also recognizes and defines exercise induced pulmonary arterial hypertension (ex-PAH), which may precede the development of resting PAH. The natural progression of PAH, especially during exercise, has not been well delineated. An exercise hemodynamic study previously showed that in normal healthy subjects the mean pulmonary pressure does not exceed 30mmHg even at maximal cardiac outputs. A prior study evaluated exercise Doppler echocardiography systemic sclerosis patients with normal resting echocardiograms, finding an abnormal response which was defined as an estimated right ventricular systolic pressure greater than 40 mmHg. In the same study, 6.6% of the patients progressed to resting PAH over the followup period of 12 months. Limited data is available regarding the prevalence of ex-PAH in systemic sclerosis using right heart catheterization.

ELIGIBILITY:
Inclusion Criteria:

1. Systemic Sclerosis diagnosed by the American College of Rheumatology consensus statement including any of the following:

   * Limited
   * Diffuse
   * Sine Scleroderma
2. Patients must be willing and able to undergo right heart catheterization with lower extremity cycle ergometry
3. Mean pulmonary artery pressure (mPAP) > 30mmHg with exercise; PCWP ≤ 15mmHg on RHC at rest
4. Men and women, ages 18 years of age or older
5. Standard adjunctive medications will be allowed concurrently in this study at the discretion of the treating pulmonologist and rheumatologist, including digoxin, diuretics, anticoagulants (e.g. warfarin), stable immunosuppression or other anti-fibrotic therapy for at least one month prior to enrollment

Exclusion Criteria:

1. Resting PAH (mPAP > 25mmHg) on right heart catheterization
2. Other known causes of PAH including prior venous thromboembolism, HIV infection, chronic liver disease with portal hypertension, left ventricular systolic dysfunction (e.g. LVEF < 40%), and congenital causes of PAH
3. Severe hepatic disease precluding the use of ambrisentan (AST/ALT ≥3x ULN).
4. Women who are pregnant or breastfeeding.
5. Concurrent therapy with a prostanoid or prostanoid analogue, PDE5 inhibitors, or enrolled in another active clinical study.
6. Use of any prostacyclin or endothelial receptor antagonist (ERA) within 30 days before study entry.
7. Bed or wheel chair bound or a baseline 6-Minute Walk distance (6MWD) less than 150 meters.
8. Childbearing capable women who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period.
9. New York Heart Association (NYHA) Classification: Class IV
10. Renal dysfunction (serum creatinine >2.5mg/dL).
11. Uncontrolled sleep apnea.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-03 (Actual); Primary Completion 2010-06 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rajeev Saggar, MD, Principal Investigator — University of California, Los Angeles; Dinesh Khanna, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- David Geffen School of Medicine, University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Saggar R, Khanna D, Shapiro S, Furst DE, Maranian P, Clements P, Abtin F, Dua S, Belperio J, Saggar R. Brief report: effect of ambrisentan treatment on exercise-induced pulmonary hypertension in systemic sclerosis: a prospective single-center, open-label pilot study. Arthritis Rheum. 2012 Dec;64(12):4072-7. doi: 10.1002/art.34614. PMID 22777623

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 15 participants were screened, and 12 were eligible and enrolled in the study
Period: Overall Study
Arm/Group | Ambrisentan
Started | 12
Completed | 11
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ambrisentan
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.6 (19.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in Exercise Pulmonary Hemodynamics From Baseline to Week 24
Description: We defined ePH (exercise PH) as an mPAP of 30 mmHg, PCWP of 18 mm Hg, and a transpulmonary gradient (TPG) of 15 mm Hg, where TPG equals mPAP minus PCWP. We defined ePVH (exercise pulmonary venous hypertension) as an mPAP of 30 mm Hg, PCWP of 18 mm Hg, and a TPG of 15 mm Hg. We defined eoPH (exercise out of proportion) as an mPAP of 30 mm Hg, PCWP of 18 mm Hg, and a TPG of 15 mm Hg (4). Our hypothesis was that SSc patients with normal exercise physiology and ePVH have a different patho-physiology compared to patients with pulmonary vascular disease (ePH and eoPH).
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Ambrisentan
Number analyzed (Participants) | 11
mmHg | 37.4 (8.3)
Statistical Analysis 1: Comparison: Ambrisentan; Whether change from baseline to 24-weeks is significantly different from zero; Test type: Other — comparison of means; p = .0008, t-test, 2 sided — significant at p<0.05; Mean Difference (Final Values) = -93.0

2. Secondary Outcome: Change in Distance Walked in Six Minutes From Baseline to 24 Week
Description: ATS guideline based assessment with known minimally clinically important difference
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Ambrisentan
Number analyzed (Participants) | 11
meters | 44.5 (10.3)
Statistical Analysis 1: Comparison: Ambrisentan; change from baseline to 24 weeks; Test type: Other; p = 0.00007, t-test, 2 sided; Mean Difference (Final Values) = 44.5

3. Secondary Outcome: Quality of Life (QOL) Based on SF36 and HAQ-DI
Description: Number of participants exceeding minimally important difference estimates on changes in quality of life as assessed by SF-36 (short form 36) quality of life index with mental and physical component scores, or by HAQ-DI (health assessment questionnaire disability index) limitations that may be related to musculoskeletal limitations
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Ambrisentan
Number analyzed (Participants) | 11
Participants | 0

4. Secondary Outcome: HAQ-DI (Health Assessment Questionnaire Disability Index)
Description: Assessing limitations that may be related to musculoskeletal limitations, the HAQ-DI assesses the difficulty a participant has had in the past week in 8 domains of daily living activities: dressing and grooming, arising, eating, walking, hygiene, reach, grip, and other activities. Each activity category consists of 2-3 items in which level of difficulty is scored from 0 to 3 with 0=no difficulty, 1=some difficulty, 2=much difficulty, and 3=unable to do. The 8 domain scores are averaged into a total HAQ-DI score ranging from 0 (no disability) to 3 (completely disabled).
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ambrisentan
Number analyzed (Participants) | 12
score on a scale | 1.12 (0.02)

5. Secondary Outcome: St. George's Respiratory Questionnaire
Description: To assess overall health, daily life, and perceived well-being in patients with underlying lung disease, the SGRQ is a health-related quality of life questionnaire divided into 3 components : symptoms, activity and impact. The total score (summed weights) can range from 0 to 100 with a lower score denoting a better health status.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ambrisentan
Number analyzed (Participants) | 12
score on a scale | 13.2 (11.7)

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Ambrisentan
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 1/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ambrisentan (N=12)
edema (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ambrisentan (N=12)
Upper respiratory symptoms (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Constipation (Gastrointestinal disorders) | 1 (1)
Joint and body pain (General disorders) | 1 (1)
Elevated liver function tests (Hepatobiliary disorders) | 1 (1)
Edema (Blood and lymphatic system disorders) | 5 (5)
Headache (General disorders) | 1 (1)
Tinea Corporis (Skin and subcutaneous tissue disorders) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1)
Bronchoalveolar carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Fecal incontinence (Gastrointestinal disorders) | 1 (1)
Pulled muscle (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes